CLINICAL TRIAL: NCT03003182
Title: A Prospective Cohort Study of Nasopharyngeal Carcinoma to Establish Prognostic Models, to Discover Toxicity Associated Predictors and to Validate Randomized Trials in Clinical Practice
Brief Title: A Study of Nasopharyngeal Carcinoma From Guangdong
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Prof., Sun Yat-sen University
Other Study IDs: 2016-FXY-098-Dept. of RT
Record Dates: First submitted 2016-12-18; First posted 2016-12-26 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- in clinical trials
- out of clinical trials

SUMMARY:
This prospective cohort study aims to establish prognostic models, to discover toxicity associated predictors and to validate randomized trials in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmed nasopharyngeal carcinoma;
* scanned by magnetic resonance imaging from calvaria vertex to clavicles before treatment;
* pretreatment Epstein-Barr virus deoxyribonucleic acid copy number is available;
* irradiated with intensity-modulated radiotherapy;

Exclusion Criteria:

* finishing anticancer therapy in two or more hospitals;
* pregnancy or lactation;
* diagnosed with other sort of cancer before or during the treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes patients with nasopharyngeal carcinoma in all stages.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3-years

SECONDARY OUTCOMES:
Number of participants with treatment-related acute adverse events as assessed by CTCAE v4.0 | 30-days

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang SS, Wu YS, Pang YJ, Xiao SM, Zhang BY, Liu ZQ, Chen EN, Zhang X, OuYang PY, Xie FY. Development and validation of radiologic scores for guiding individualized induction chemotherapy in T3N1M0 nasopharyngeal carcinoma. Eur Radiol. 2022 Jun;32(6):3649-3660. doi: 10.1007/s00330-021-08460-1. Epub 2022 Jan 6. PMID 34989842